CLINICAL TRIAL: NCT01874795
Title: Effect of Ganglionar Transcutaneous Electrical Nerve Stimulation on Central Arterial Pressure in Healthy Young Population
Brief Title: Effect of Ganglionar Electrical Stimulation on Central Arterial Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Gerson Cipriano Jr, PhD, University of Brasilia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 071/2011
Record Dates: First submitted 2012-07-11; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Heart Failure; Chagas Disease
Keywords: Autonomic Nervous System; Neuromodulation; Exercise; Pulmonary oxygen kinetics; Oxygen uptake
MeSH Terms: conditions — Heart Failure; Chagas Disease; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ganglionar Electrical Stimulation (Experimental): TENS intervention consisted of continuous flow, symmetrical and rectangular TENS biphasic pulses. The frequency ofstimulation was 80 Hz and the pulse duration was 150 μs, with the intensity in adjusted to the point of muscle contraction.
  Interventions: Device: TENS
- Placebo (Sham Comparator): The frequency of stimulation was 80 Hz and the pulse duration was 150 μs, equipment did not provide stimulation current.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: TENS — Adhesive electrodes (MultiStick®, USA) were placed on each side, about 3 cm to the right and left of midline vertebral process, at C7 (Channel 1) and T4 (Channel 2).
  Other Names: Ganglionar electrical stimulation
  Arms: Ganglionar Electrical Stimulation
Device: Placebo — The frequency of stimulation was 80 Hz and the pulse duration was 150 μs, equipment did not provide stimulation current.
  Arms: Placebo

SUMMARY:
This study will evaluate the applications of ganglionar electrical stimulation in patients with Chagas Disease and Ischemic Heart Failure patients.

DETAILED DESCRIPTION:
A Crossover Randomized Controlled Study will be developed with 3 groups: Healthy Older, Ischemic Heart Failure and Chagas Disease. This individuals will be randomized in two groups: TENS and placebo (same stimulus without electrical output) with 48 hrs between the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic and Chagas disease previously diagnosticated
* Age above 40 years old

Exclusion Criteria:

* No vascular disease
* No recent surgery
* No recent infections

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
tonometry | participants will be followed for the duration of myostimulation protocol, an expected average of 5 weeks
  Applanation tonometry (AT) accurately reflects arterial stiffness method and has demonstrated a strong correlation with ventricular-vascular coupling. Increased arterial stiffness and wave reflection have also been reported in patients with systolic and diastolic HF.

SECONDARY OUTCOMES:
Cardiorespiratory Evaluation | participants will be followed for the duration of myostimulation protocol, an expected average of 5 weeks
  Cardiopulmonary exercise testing (CPX) is a highly reliable and valid approach to assessing aerobic performance. It is a well-accepted assessment technique in the HF population with American and European associations endorsing its use. CPX is most often performed on a treadmill or cycle ergometer using ramping protocols and the addition of ventilatory expired gas analysis to the standard exercise test enables measurement of oxygen consumption (VO2), carbon dioxide production (VCO2) and minute ventilation (VE) over time. Moreover, CPX provides a host of variables that are predictive of adverse events in HF patients, including peak VO2, the VE/VCO2 slope and the oxygen uptake efficiency slope (OUES).

CONTACTS AND LOCATIONS:
Overall Officials: Gerson C junior, PhD, Principal Investigator — University of Brasilia; Gaspar R Chiappa, ScD, Principal Investigator — University Federal of Rio Grande do Sul
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Cipriano G Jr, de Camargo Carvalho AC, Bernardelli GF, Tayar Peres PA. Short-term transcutaneous electrical nerve stimulation after cardiac surgery: effect on pain, pulmonary function and electrical muscle activity. Interact Cardiovasc Thorac Surg. 2008 Aug;7(4):539-43. doi: 10.1510/icvts.2007.168542. Epub 2008 Apr 16. PMID 18417519
- [Background] Chiappa GR, Borghi-Silva A, Ferreira LF, Carrascosa C, Oliveira CC, Maia J, Gimenes AC, Queiroga F Jr, Berton D, Ferreira EM, Nery LE, Neder JA. Kinetics of muscle deoxygenation are accelerated at the onset of heavy-intensity exercise in patients with COPD: relationship to central cardiovascular dynamics. J Appl Physiol (1985). 2008 May;104(5):1341-50. doi: 10.1152/japplphysiol.01364.2007. Epub 2008 Mar 20. PMID 18356477
- [Background] Vieira PJ, Ribeiro JP, Cipriano G Jr, Umpierre D, Cahalin LP, Moraes RS, Chiappa GR. Effect of transcutaneous electrical nerve stimulation on muscle metaboreflex in healthy young and older subjects. Eur J Appl Physiol. 2012 Apr;112(4):1327-34. doi: 10.1007/s00421-011-2084-z. Epub 2011 Jul 28. PMID 21796410